CLINICAL TRIAL: NCT04639518
Title: Growth and Safety of Two Partially-hydrolyzed Feeding Systems for Preterm Infants: a Multi-centered, Open-label Clinical Trial
Brief Title: Growth and Safety of Two Partially-hydrolyzed Feeding Systems for Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 18.09.INF
Record Dates: First submitted 2020-10-22; First posted 2020-11-20 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Pre-term Infant
MeSH Terms: interventions — Health Maintenance Organizations

STUDY DESIGN:
Intervention Model Description: Two sequential sub-studies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sub-study 1 (Experimental): Pre-term formulas with HMO
  Interventions: Other: Preterm formulas with HMO
- Sub-study 2 (Experimental): Pre-term formulas without HMO
  Interventions: Other: Preterm formulas without HMO

INTERVENTIONS:
Other: Preterm formulas with HMO — Preterm infants will receive Stage 1 formula as soon as possible after birth until when 1.8 kg of body weight is achieved. Preterm infants will receive Stage 2 preterm formula from when 1.8 kg of body weight is achieved until 2 months after hospital discharge.
  Arms: Sub-study 1
Other: Preterm formulas without HMO — Preterm infants will receive Stage 1 formula as soon as possible after birth until when 1.8 kg of body weight is achieved. Preterm infants will receive Stage 2 preterm formula from when 1.8 kg of body weight is achieved until 2 months after hospital discharge.
  Arms: Sub-study 2

SUMMARY:
This is an open-label trial consisting of two sub-studies to be conducted sequentially with the purpose of evaluating the safety and suitability of a two feeding systems in pre-term infants (one containing HMOs and one without HMOs).

DETAILED DESCRIPTION:
This is a multi-center, open-label trial to be conducted in up to 70 pre-term infants in order to evaluate the safety and suitability of two feeding systems as they would typically be used in the neonatal care unit. Growth (in comparison to recommended growth goals), feeding tolerance, biochemical parameters, and adverse event reporting will be evaluated.

The two feeding systems will be tested in two sub-studies to be conducted sequentially: sub-study 1 will evaluate a two-staged feeding system with HMOs in up to 35 pre-term infants; sub-study 2 will evaluate a two-staged feeding system without HMOs in up to 35 pre-term infants.

A follow up period from 12 to 24 months have been added to the study protocol, to assess the neurocognitive development of the subjects during this period.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent has been obtained from one or both parent(s) /legally acceptable representative (LAR) in accordance with local regulation.
2. Infants' birth weight ≤1500 g and AGA.
3. Infant's gestational age < 37 weeks.
4. Infant is clinically stable and does not have deteriorating respiratory function after birth.
5. Infant is eligible to start experimental formula after 24 hours of trophic feeding, but still within the first 10 days (≤240 hours) of life.

Exclusion Criteria:

1. Parent(s) not willing / not able to comply with the requirements of study protocol.
2. Infant is experiencing early onset sepsis.
3. Major congenital or chromosomal abnormality known to affect growth.
4. Liver failure.
5. Peri-/intra-ventricular haemorrhage (grade 3-4 in Papille classification).
6. Infant who has siblings with diagnosed allergies or intolerances to lactose or cow's milk.
7. Infant's participation in another interventional clinical trial.
8. Infant has already achieved FEF prior to enrolment, using the definition accepted by Neonatal Unit as per standard practice (150 mL/kg/day).

Max Age: 10 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2020-09-10 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2025-04-28 (Actual)

PRIMARY OUTCOMES:
Growth | From FEF Day 1 to when infant reaches 1800 g (on average between 4 to 6 weeks after birth) or hospital discharge (on average 7 weeks after birth), whichever comes earlier
  Weight-adjusted weight gain (g/kg/day)

SECONDARY OUTCOMES:
Weight at other time points | From Pre-FEF Day 1 to FEF Day 1, and then weekly from FEF Day 1 until hospital discharge (on average 7 weeks after birth), at 30- and 60-days PD, and at 12, 18, and 24 months
  Changes in weight gain (g/day and g/kg/day)
Other growth parameter (length) | From Pre-FEF Day 1 to hospital discharge (on average 7 weeks after birth), at 30- and 60-days PD, and at 12, 18, and 24 months
  Change in length (cm/week)
Other growth parameter (head circumference) | From Pre-FEF Day 1 to hospital discharge (on average 7 weeks after birth), at 30- and 60-days PD, and at 12, 18, and 24 months
  Change in head circumference (cm/week)
Anthropometric z-scores for weight, length and head circumference | From Pre-FEF Day 1 to hospital discharge (on average 7 weeks after birth), at 30- and 60-days PD, and at 12, 18, and 24 months
  Corresponding z-scores and changes in z-scores expressed using Fenton growth chart will be analyzed
Feeding intake at neonatal unit | Baseline + weekly over 3 consecutive days starting on pre-FEF Day1 + weekly over 3 consecutive days starting on FEF Day1 until Neonatal Unit Discharge (on average 7 weeks after birth)
  Neonatal unit feeding questionnaire capturing timing, type, rate and amount of feeding (parenteral & enteral), gastric residual volumes, number of missed feedings
Stool frequency at neonatal unit | Weekly between FEF Day 1 and hospital discharge (on average 7 weeks after birth)
  Stool frequency (range from 0-20 times a day) collected via neonatal unit questionnaire
Stool consistency at neonatal unit | Weekly between FEF Day 1 and hospital discharge (on average 7 weeks after birth)
  Stool consistency (watery, mushy soft, runny, formed, hard) collected via neonatal unit questionnaire
Bloody stools at neonatal unit | Weekly between FEF Day 1 and hospital discharge (on average 7 weeks after birth)
  Bloody stools (yes or no) collected via neonatal unit questionnaire
GI symptoms at neonatal unit | Weekly between FEF Day 1 and hospital discharge (on average 7 weeks after birth)
  GI symptoms (incidence of abdominal distention, regurgitation, spitting and vomiting) collected via neonatal unit questionnaire
Feeding intake after discharge | 3 consecutive days just prior to the 30-day PD and 60-day PD visits
  Parent-reported 3-Day Intake Diary capturing the total number of bottles of formula and approximate volumes consumed per day
Stool frequency after discharge | 3 consecutive days just prior to the 30-day PD and 60-day PD visits
  Stool frequency captured via parent-reported 3-Day Intake Diary
Stool consistency after discharge | 3 consecutive days just prior to the 30-day PD and 60-day PD visits
  Stool frequency captured via parent-reported 3-Day Intake Diary
GI symptoms after discharge | 3 consecutive days just prior to the 30-day PD and 60-day PD visits
  GI symptoms (such as presence of stomach ballooning, bloody stools, regurgitation, spitting-up and vomiting) captured via parent-reported 3-Day Intake Diary
GI-related behaviors after discharge | 3 consecutive days just prior to the 30-day PD and 60-day PD visits
  GI-related behaviors (such as crying and sleep quality) captured via parent-reported 3-Day Intake Diary
Serum biomarkers for protein status | At Baseline (if possible), pre-FEF Day 1, then weekly pre-FEF Days 7, 14, etc. and FEF Day 1, then weekly on FEF Days 7, 14, 21, until Neonatal Unit Discharge, and at 60 days PD
  Serum albumin and blood urea nitrogen (BUN)
Serum biomarkers for bone health | At Baseline (if possible), pre-FEF Day 1, then weekly pre-FEF Days 7, 14, etc. and FEF Day 1, then weekly on FEF Days 7, 14, 21, until Neonatal Unit Discharge, and at 60 days PD
  Serum P, alkaline phosphatase, calcium and creatinine
Urine biomarkers for bone health | At Baseline (if possible), pre-FEF Day 1, then weekly pre-FEF Days 7, 14, etc. and FEF Day 1, then weekly on FEF Days 7, 14, 21, until Neonatal Unit Discharge, and at 60 days PD
  Urinary Ca, P and creatinine
Vitamin D | FEF Day 1, Neonatal Unit Discharge and at 60 days PD
  Vitamin D
Fecal microbiota | Baseline, FEF Day 1, then weekly on FEF Days 7, 14, 21, until Neonatal Unit Discharge, at 30 day-PD and 60 days PD
  Fecal microbiota composition, diversity and metabolism markers (SCFAs)
Fecal markers for gut health / maturation and immune status | Baseline (if feasible), FEF Day 1, Day 21, Neonatal Unit Discharge, 30 day-PD and 60 day-PD
  Fecal levels of calprotectin, alpha 1 antitrypsin, pancreatic elastase (i.e. chymotrypsin-like elastase family, member 3B (CELA3B)), Human beta-defensin 2 (HBD2) and secretory IgA
Urine markers for gut health / maturation and immune status | Baseline (if feasible), FEF Day 1, Day 21, Neonatal Unit Discharge, 30 day-PD and 60 day-PD
  Urinary level (spot urine sample) of intestinal fatty acid binding protein (iFABP)
AE reporting | From the time the mother has consented to the infant's participation in the study until the 60 days PD visit
  Number of AEs through investigator-confirmed AE reporting
Bayley-III scores | At 12, 18, and 24 months
  Bayley scales of Infants and Toddler development - 3rd edition
Developmental Milestone scores | At 12, 18, and 24 months
  Parent-reported achievements of specific-age appropriate milestones (yes/no reponses to child performing specific milestones or not)
Child temperament scores | At 12, 18, and 24 months
  Parent-reported child temperament questionnaire
Number of healthcare usage | At 12, 18, and 24 months
  Retrospective paret-reported recall of the number of healthcare usage and hospitalizations
Feeding patterns | At 12, 18, and 24 months
  Feeding practice outcomes collected retrospectively at each visit via a parent-reported questionnaire related to breastfeeding duration, prevalence of formula feeding, and age at initiation of complementary feeding

CONTACTS AND LOCATIONS:
Locations (4):
- Klinikum Nuernberg, Nuremberg, Germany
- Klinika Neonatologii, Szpital Uniwersyteck, Bydgoszcz, Poland
- Slovakia (2):
  - Univerzitna nemocnica Martin, Martin
  - Fakultna nemocnica s poliklinikou Nove Zamky, Nové Zámky

IPD SHARING:
Plan to Share IPD: No